CLINICAL TRIAL: NCT07398729
Title: The Effects of Short-term Motivational Factors and Calisthenic Exercise on Blood Cortisol Levels, and Symptoms of Depression, Anxiety, and Stress in Young Adults
Brief Title: Physiological and Psychological Effects
Acronym: DASS21-CORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bingol University (Other)
Responsible Party: Principal Investigator, Mehmet Kaplan, Asst. Prof., Bingol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: BAP-SHMYO.2025.001; BAP-SHMYO.2025.001 (Other Grant/Funding Number: Bingol University)
Record Dates: First submitted 2026-01-25; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Healthy Young Adults
Keywords: Anxiety; Calisthenic exercise; Cortisol; Depression; Motivational factors; Stress; Young adult
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: This study is a three-arm, randomised controlled trial.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): No intervention was applied to this group.
- MF group (Experimental): Only motivational factors were applied to this group. As motivational factors, participants performed diaphragmatic breathing exercises and stretching exercises in groups.
  Interventions: Other: Motivational factors
- MF+CE group (Experimental): Motivational factors and calisthenic exercises were applied to this group. First, motivational factors were implemented in groups, followed by calisthenic exercises.
  Interventions: Other: Calisthenic exercise and Motivational factors; Other: Motivational factors

INTERVENTIONS:
Other: Calisthenic exercise and Motivational factors — Following a 15-minute motivational factors intervention, a 30-minute calisthenic exercise program was implemented.
  Other Names: CE and MF
  Arms: MF+CE group
Other: Motivational factors — A 15-minute motivational factors intervention was applied.
  Arms: MF group; MF+CE group

SUMMARY:
Stress-related mental health problems such as depression, anxiety, and stress are common among young adults and are often linked to both psychological and physiological changes in the body. One of the key biological markers of stress is cortisol, a hormone released in response to stress. Elevated cortisol levels over time may negatively affect both mental and physical health. Although regular physical activity and relaxation-based approaches are known to reduce stress, it is not yet clear whether short-term, easily applicable interventions can produce measurable benefits, especially when motivational strategies and exercise are combined.

The purpose of this study is to evaluate the effects of short-term motivational factors and a single session of calisthenic exercise on blood cortisol levels and symptoms of depression, anxiety, and stress in young adults. Motivational factors in this study include group-based activities, diaphragmatic breathing, and stretching exercises, which are designed to increase engagement and relaxation without requiring intense physical effort. Calisthenic exercise refers to bodyweight-based movements that can be performed without special equipment and are accessible to most individuals.

This randomized controlled trial compares three groups: one group receiving motivational factors followed by a single session of calisthenic exercise, a second group receiving motivational factors only, and a control group receiving no intervention. By measuring blood cortisol levels and self-reported symptoms of depression, anxiety, and stress before and after the intervention, the study aims to determine whether these short-term interventions can lead to meaningful psychological and physiological improvements.

The main question this study seeks to answer is whether a brief, single-session intervention combining motivational strategies and calisthenic exercise is more effective than motivational strategies alone or no intervention in reducing stress hormone levels and psychological distress in young adults. Additionally, the study explores whether lifestyle and sociodemographic factors, such as exercise habits, sleep patterns, and perceived economic status, are associated with cortisol levels.

The findings of this study may help identify simple, low-cost, and time-efficient approaches that can be used to support stress management and mental well-being in young adult populations, particularly in university settings.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who voluntarily agreed to participate.
* Individuals aged between 18 and 25 years.
* Individuals who had not engaged in regular exercise (at least three days per week) within the past six months.
* Individuals with no diagnosed psychiatric disorder.
* Individuals with no chronic health condition.
* Individuals who did not use any substances.

Exclusion Criteria:

* Individuals who did not agree to participate in the study.
* Individuals who completed the baseline (pre-intervention) assessment but did not complete the post-intervention assessment.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2025-07-02 (Actual); Primary Completion 2025-11-19 (Actual); Study Completion 2026-01-20 (Actual)

PRIMARY OUTCOMES:
DASS-21 | Immediately before and immediately after the single 45-minute exercise session
  It is scored between 0 and 63. Higher scores indicate higher levels of depression, anxiety, and stress.
Cortisol | Immediately before the exercise session and 20 minutes after completion of the single exercise session
  Blood cortisol concentration will be measured in µg/dL using a standardized laboratory assay.
  A value of 17 µg/dL is considered a commonly used reference threshold, with values above this level generally indicating higher physiological stress and values below this level indicating lower physiological stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Bingöl University, Merkez, Bingöl, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the dataset contains sensitive personal and biological information, and data sharing was not included in the informed consent obtained from participants.